CLINICAL TRIAL: NCT06063057
Title: Inactivated Bivalent Enterovirus Vaccine Phase I/II Clinical Trial: Open-Label Observation in Healthy Adults and Children, and Randomized, Double-Blind, Controlled Clinical Trial in Children
Brief Title: Inactivated Bivalent Enterovirus Vaccine (Vero Cell) Phase I/II Clinical Trial
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-EV71/CA16-1001
Record Dates: First submitted 2023-09-15; First posted 2023-10-02 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hand, Foot and Mouth Disease; Herpangina
Keywords: Inactivated enterovirus vaccine; Bivalent enterovirus vaccine
MeSH Terms: conditions — Hand, Foot and Mouth Disease; Herpangina

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- low-dose experimental group (Experimental): phase Ⅰ: 18~59 years old,6~12 years old,6~71 months old; phase Ⅱ：6~71 months old
  Interventions: Biological: low dose Bivalent Enterovirus Vaccine (Vero Cell), Inactivated
- medium-dose experimental group (Experimental): phase Ⅰ: 18~59 years old,6~12 years old,6~71 months old; phase Ⅱ：6~71 months old
  Interventions: Biological: medium dose Bivalent Enterovirus Vaccine (Vero Cell), Inactivated
- high-dose experimental group (Experimental): phase Ⅰ: 18~59 years old,6~12 years old,6~71 months old; phase Ⅱ：6~71 months old
  Interventions: Biological: high dose Bivalent Enterovirus Vaccine (Vero Cell), Inactivated
- Active control group (Active Comparator): phase Ⅰ: 6~71 months old; phase Ⅱ：6~71 months old
  Interventions: Biological: Enterovirus type EV71 vaccine (Vero cell), Inactivated

INTERVENTIONS:
Biological: low dose Bivalent Enterovirus Vaccine (Vero Cell), Inactivated — Bivalent Enterovirus Vaccine (Vero Cell), Inactivated antigen content: EV71 480 U-CA16 600 SU/0.5 ml
  Arms: low-dose experimental group
Biological: medium dose Bivalent Enterovirus Vaccine (Vero Cell), Inactivated — Bivalent Enterovirus Vaccine (Vero Cell), Inactivated antigen content: EV71 960 U-CA16 600 SU/0.5 ml
  Arms: medium-dose experimental group
Biological: high dose Bivalent Enterovirus Vaccine (Vero Cell), Inactivated — Bivalent Enterovirus Vaccine (Vero Cell), Inactivated antigen content: EV71 1920U-CA16 1200SU/0.5ml
  Arms: high-dose experimental group
Biological: Enterovirus type EV71 vaccine (Vero cell), Inactivated — Enterovirus type EV71 vaccine (Vero cell), Inactivated (Sinovac)
  Arms: Active control group

SUMMARY:
The Phase I clinical trial is divided into two parts. The first part uses an open-label design, while the second part uses a randomized, double-blind, and controlled design. The goal of this clinical trial is to evaluate the tolerability and safety of a bivalent (EV71/CA16, Enterovirus 71/Coxsackievirus A16) inactivated enterovirus vaccine (Vero cell) developed by Sinovac. The vaccine will be administered to healthy adults, children aged 6 to 12 years, and children aged 6 to 71 months.

The Phase II clinical trial will also use a randomized, double-blind, and controlled design to evaluate the safety and immunogenicity of the same bivalent inactivated enterovirus vaccine (Vero cell) developed by Sinovac. This trial will involve healthy children aged 6 to 71 months.

DETAILED DESCRIPTION:
For phase I clinical trial:

The first part of the trial plans to recruit thirty-six healthy adults aged 18-59 years and thirty-six children aged 6-12 years, with twelve participants in each of the low-dose (EV71 480 U-CA16 600 SU/0.5 ml), medium-dose (EV71 960 U-CA16 600 SU/0.5 ml), and high-dose (EV71 1920U-CA16 1200SU/0.5ml) experimental groups. The participants will receive two doses of the experimental vaccine according to a 0-1-month schedule, with adults vaccinated before children.

The second part of the trial plans to recruit seventy-two healthy children aged 6-71 months, with each dose group having twelve participants in the 6-23 months and 24-71 months age groups. The participants will receive two doses of the experimental vaccine according to a 0-1-month schedule, with each dose group being randomized, double-blind, and positive-controlled. The vaccine will be compared to a control (EV71 vaccine) at each dose level.

The dose escalation principle within each age group is from low to high doses: After completing the first dose of the lower dose stage, a safety observation period of 0-7 days will be conducted to confirm safety based on adverse event occurrence and blood routine, blood biochemistry, and urine routine tests (if any) before proceeding to the higher dose stage. The sequential enrollment principle between different age groups is from adults and children aged 6-12 years to children aged 6-71 months. After the first dose of each dose group is administered to adults, children aged 6-12 years in the same dose group can be enrolled only after a safety observation period of 0-7 days confirms safety. After completing the second dose of the medium-dose group in adults, vaccination of children aged 6-71 months can begin.

Participants in the adult and children aged 6-12 years groups will have approximately 5.5 mL of blood (2.0 mL anticoagulated blood and 3.5 mL non-anticoagulated blood) and about 2-10 mL of urine samples collected before and on day three after each dose for blood routine, blood biochemistry, and urine routine tests to evaluate vaccine safety. Only participants aged 24-71 months in the second stage of the trial will undergo these tests before the first dose. Whether participants aged 24-71 months to conduct tests on days 3 (Visit2), 30 (Visit5), and 33 (Visit6) will depend on the relevant test results in the children aged 6-12 years group. If 10% of participants in each dose stage of the children aged 6-12 years group have abnormal test results related to the vaccine that is clinically significant after the first dose, blood and urine samples will be collected from corresponding dose stage participants aged 24-71 months on days 3 (Visit2), 30 (Visit5), and 33 (Visit6).

For phase II clinical trial:

A total of six hundred children aged 6-71 months will be recruited, including 360 children aged 6-23 months and 240 children aged 24-71 months. The participants will be randomly allocated to the low-dose (EV71 480U-CA16 600SU/0.5ml), medium-dose (EV71 960U-CA16 600SU/0.5ml), high-dose (EV71 1920U-CA16 1200SU/0.5ml) experimental groups and control group (EV71 vaccine) in a 1:1:1:1 ratio.

Participants will be given two doses of either the experimental or control vaccine, administered one month apart.

During phase II of the trial, all participants will undergo blood collection on three different days: day zero, day sixty, and day 210 after vaccination. The collection will involve approximately 3.0 mL of venous blood to be separated into serum for EV71 and CA16 neutralizing antibodies assays. These assays will help evaluate the immunogenicity and immune persistence of the vaccine.

All participants in phases I/II will be observed for immediate reactions within 30 minutes after each dose, and adverse events (AEs) will be collected for the first seven days after each dose and non-solicited AEs for the first 30 days after each dose. Serious adverse events (SAEs) will be monitored from the start of vaccination until six months after completion of the vaccination course. In phase I, pregnancy events within three months (120 days) after vaccination will be collected based on self-report.

Once safety data for all participants has been obtained for 30 days after completing the vaccination course in phase I, the investigators will seek ethics approval. If the safety results are deemed satisfactory and approved by the ethics committee, the investigators will move forward to phase II clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants aged 18-59 years, 6-12 years, and 6-71 months.
* Participants and/or their guardians can understand and voluntarily sign the informed consent form (participants aged 8-12 years require dual signatures from both participants and their guardians).
* Willing and able to comply with all visit schedules, sample collection, vaccine administration, and other trial procedures.
* Provide legal identification of the participants and/or their guardians.

Exclusion Criteria:

* History of hand, foot, and mouth disease or EV71 vaccination.
* Known severe allergy to the vaccine or vaccine components, such as urticaria, respiratory distress, and angioedema.
* Congenital abnormalities or developmental disorders, genetic defects (such as Down syndrome, thalassemia, or G6PD deficiency), severe malnutrition, etc.
* Based on medical history and physical examination, the presence of severe chronic diseases, severe cardiovascular diseases, uncontrolled hypertension or diabetes, liver or kidney diseases, etc.
* Based on medical history and physical examination, the presence of autoimmune diseases, immunodeficiency diseases, and/or blood diseases (including but not limited to systemic lupus erythematosus, ankylosing spondylitis, thyroidectomy, autoimmune thyroid disease, any form of malignancy, asplenia, functional asplenia).
* Based on medical history and physical examination, abnormal coagulation function (such as coagulation factor deficiency, coagulation disorders, platelet abnormalities) or obvious bruising or bleeding disorders.
* Based on medical history and physical examination, the presence of severe neurological diseases (epilepsy, convulsions, or seizures), mental illness, or corresponding family history.
* Long-term use (more than 14 days) of corticosteroids or other immunosuppressive agents (excluding corticosteroid sprays for allergic rhinitis and surface corticosteroid treatment for acute non-complicated dermatitis) or cytotoxic therapy or planning to receive such treatment during the trial.
* History of long-term alcohol abuse or drug abuse.
* Females who are breastfeeding, pregnant, or planning to become pregnant within 90 days, or females with positive pregnancy test results. Note: male participants whose spouse plans to become pregnant within 90 days are also included.
* Received immunoglobulin and/or other blood products in the past 3 months or planning to receive such treatment during the trial.
* Received other investigational drugs or vaccines within the past 30 days or planning to receive such drugs or vaccines during the trial.
* Vaccinated with attenuated live vaccines within the past 14 days or subunit or inactivated vaccines within the past 7 days.
* Suspected or confirmed fever within 72 hours before vaccination or axillary temperature >37.0℃ on the day of vaccination.
* Clinical laboratory testing shows laboratory abnormalities beyond the reference range and with clinical significance (applicable only to Phase I clinical trials for adults/6-12-year-old children/24-71-month-old children):

A. Complete blood count: white blood cell count, hemoglobin, platelet count.B. Blood biochemistry: alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (TBIL), creatinine (CR), fasting blood glucose (Glu).C. Urine routine: urine protein (PRO).

* Any acute illness (with or without fever) or exacerbation of chronic illness within the past 7 days.
* According to the investigator's judgment, there are any other factors that make the participant unsuitable for participation in the clinical trial.

Ages: 6 Months to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 744 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Phase Ⅰ: Based on adverse events, evaluate the safety of the trial vaccine among participants in different age groups | 30 days
  the incidence rates of adverse reactions from the start of vaccination to 30 days after the end of the entire vaccination course
Phase Ⅱ: Evaluate the immunogenicity of the trial vaccine in the target population. | 30 days
  The seroconversion rate of EV71 and CA16 neutralizing antibodies in children aged 6-71 months 30 days after the end of the entire vaccination course.

SECONDARY OUTCOMES:
Phase Ⅰ: Based on adverse events, evaluate the safety of the trial vaccine among participants in different age groups. | 7 days
  - The incidence rate of adverse reactions from 0-7 days after each dose.
Phase Ⅰ: Based on adverse events, evaluate the safety of the trial vaccine among participants in different age groups. | 6 months
  - The incidence rate of serious adverse events from the start of vaccination to 6 months after the end of the entire vaccination course.
Phase Ⅰ: Based on laboratory abnormalities, evaluate the safety of the trial vaccine among participants in different age groups. | 3 days
  -The incidence rate of clinically significant abnormal blood biochemistry, blood routine, and urine routine indexes within 3 days after each dose.
Phase Ⅱ: Evaluate other immunogenicity indicators of the trial vaccine. | 30 days
  -The seropositive rates of EV71 and CA16 neutralizing antibodies 30 days after the end of the entire vaccination course.
Phase Ⅱ: Evaluate other immunogenicity indicators of the trial vaccine. | 30 days
  -The GMTs (Geometric Mean Titers) of EV71 and CA16 neutralizing antibodies 30 days after the end of the entire vaccination course.
Phase Ⅱ: Evaluate other immunogenicity indicators of the trial vaccine. | 30 days
  -The GMFRs (Geometric Mean Fold Rise) of EV71 and CA16 neutralizing antibodies 30 days after the end of the entire vaccination course.
Phase Ⅱ: Based on adverse events, evaluate the safety of the trial vaccine. | 30 days
  -The incidence rate of adverse reactions from the start of vaccination to 30 days after the end of the entire vaccination course.
Phase Ⅱ: Based on adverse events, evaluate the safety of the trial vaccine. | 7 days
  -The incidence rate of adverse reactions from 0-7 days after each dose.
Phase Ⅱ: Based on adverse events, evaluate the safety of the trial vaccine. | 6 months
  -The incidence rate of SAEs from the start of vaccination to 6 months after the end of the entire vaccination course.
Phase Ⅱ: Evaluate the immune persistence of the trial vaccine. | 6 months
  -The seropositive rates of neutralizing antibodies against EV71 and CA16 6 months after the vaccination course.
Phase Ⅱ: Evaluate the immune persistence of the trial vaccine. | 6 months
  -The seropositive rates of EV71, and CA16 neutralizing antibodies 6 months after the end of the entire vaccination course.
Phase Ⅱ: Evaluate the immune persistence of the trial vaccine. | 6 months
  -The GMTs of EV71, and CA16 neutralizing antibodies 6 months after the end of the entire vaccination course.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Yan, Principal Investigator — Yunnan Provincial Center for Disease Control and Prevention
Locations (1):
- Dayao County Center for Disease Control and Prevention, Chuxiong, Yunnan, China